CLINICAL TRIAL: NCT04722744
Title: Marginal Bone Changes of CAD/CAM Implant Supported Screw-retained Metal Frameworks Based on Actual Versus Screwmented Ones Based on Virtual Implant Position: A Randomized Clinical Stud
Brief Title: Marginal Bone Changes of CAD/CAM Implant Supported Screw-retained and Screw-mented Metal Frameworks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Magdy Ibrahim, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 101120
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Patient Satisfaction; Bone Loss
MeSH Terms: conditions — Patient Satisfaction; Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- screwmented metal frameworks based on virtual implant position. (Experimental): this group will receive a CAD CAM restoration based on virtually planned implant position.
  Interventions: Procedure: screwmented metal frameworks
- screw-retained metal frameworks based on actual implant position. (Active Comparator): this group will receive screw retained CAD CAM restoration based on actual implant position using conventional open tray impression.
  Interventions: Procedure: screwmented metal frameworks

INTERVENTIONS:
Procedure: screwmented metal frameworks — Intervention group: in which the edentulous area will be restored with 3-implant, screwmented CAD/CAM frameworks constructed based on planned implant positions

SUMMARY:
compare CAD/CAM implant supported screw-retained metal frameworks based on actual versus screw-mented ones based on virtual implant position regarding marginal bone changes.

DETAILED DESCRIPTION:
patients with at least three missing teeth will be recruited and randomly assigned into two parallel groups. both groups will receive three implants based on planned implant positions and then one group will receive screw retained CAD CAM restoration with conventional impression technique while the second group will receive screw-mented CAD CAM restoration based on planned implant positions.

ELIGIBILITY:
Inclusion Criteria:

* Kennedy class I, II Or IV cases.
* Opposing completely dentulous, fully or partially restored dentition.
* Good oral hygiene.
* The patient should have bone for implants, minimum bone height 10 mm and minimum bone diameter should be 6 mm.
* Adequate inter arch space for restoration 15mm or more.
* Adult patients age ≥18 years

Exclusion Criteria:

* any medical disorder that could complicate surgical phase or affect osteointegration. Radiation chemotherapy.
* smokers more than 10/daily.
* Uncooperative patients.
* Patients with Para-functional habits
* Patients with severe periodontal diseases.
* Patients with limited mouth opening.
* Presence of intraoral pathological lesions.
* Diabetic (HbA1c >7.5%).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
marginal bone changes. | 6 months
  Using long cone paralleling technique , RINN XCP and Digora (digital periapical radiographs for standardization. the bone loss is measured in mm

SECONDARY OUTCOMES:
Patient satisfaction | 6 months
  Patient satisfaction questionnaire using Visual Analogue Scale (VAS) scale, from 0-100, where 0 is the worst meaning that patient is not satisfied and 100 is the highest satisfaction meaning the patient is totally satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Azza Hussein, PhD, Study Chair — Professor of Prosthodontics; Mohamed ElKhashab, PhD, Study Director — Lecturer of prosthodontics; Iman Radi, PhD, Study Director — Professor of Prosthodontics
Locations (1):
- Faculty of Dentistry, Cairo, Manial, Egypt